CLINICAL TRIAL: NCT01287234
Title: Atrio-Ventricular Delay Optimization in Patients Implanted With a Cardiac Resynchronization Device Using Echocardiography Versus the SonR Signal: A Pilot Study
Brief Title: Atrio-Ventricular (AV) Delay Optimization Using Echocardiography Versus the SonR Signal
Acronym: SonR Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Piedmont Healthcare (Other)
Collaborators: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SonR Pilot
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Patients (Other): All patients will have an echocardiogram and SonR sensor readings completed.
  Interventions: Other: Echocardiogram/SonR

INTERVENTIONS:
Other: Echocardiogram/SonR — All patients will have an echocardiograph and SonR sensor readings

SUMMARY:
The purpose of this study is to evaluate an external device (SonR sensor) that is capable of detecting sounds created by the heart (SonR signal). Based on the sounds created by the heart and recorded by the SonR sensor, optimal timing settings for the cardiac resynchronization therapy defibrillator (CRT-D) device may be determined. The investigators will then compare the timing settings suggested by SonR to the settings suggested from the echocardiogram. The objective of this study is to determine if differences exist between these different methods of timing the contractions of the top and bottom chambers of the heart and if the SonR signal is able to produce results similar to those of an echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with any current Food and Drug Administration (FDA) approved CRT- D device and leads for 30 days or patients indicated for AV optimization
* ≥18 years of age
* Ability and willingness to provide written informed consent and HIPAA authorization

Exclusion Criteria:

* Chronic Atrial Fibrillation
* Heart Failure decompensation event within two weeks of enrollment
* Hypertrophic Obstructive Cardiomyopathy
* Patient currently enrolled in another ongoing clinical trial
* Pregnancy
* Less than 18 years of age
* Inability or unwillingness to provide written informed consent and HIPAA authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Optimal blood flow method | 3 months
  To determine the best method of timing the contractions of the top and bottom chambers of the heart by using echocardiography versus using signals of the external SonR sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Dan, MD, Principal Investigator — Piedmont Heart Institute
Locations (1):
- Piedmont Heart Institute, Atlanta, Georgia, United States